CLINICAL TRIAL: NCT04041986
Title: Transcranial Direct Current Stimulation Investigations of Language Processing in Aphasia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 811842
Record Dates: First submitted 2019-07-11; First posted 2019-08-01 (Actual); Last update posted 2019-08-01 (Actual); Status verified 2019-07

CONDITIONS: Aphasia
Keywords: stroke; non-invasive brain stimulation; transcranial direct current stimulation (tDCS)
MeSH Terms: conditions — Aphasia; Stroke | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: This is an incomplete crossover design where subjects randomized to the real tDCS group will end their participation but subjects randomized to the sham tDCS group will crossover into the real tDCS group.
Who Masked: Participant
Masking Description: Participants will be blinded to which tDCS group (real or sham) they are initially enrolled in; however, since only the sham group crosses over this will signal to subject that they are now getting real stimulation.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Site-Finding (Experimental): Each subject will receive anodal, cathodal, and sham stimulation to both the ipsilesional and contralesional hemispheres in a series of six sessions (one condition per session), each separated by at least two days. During anodal and cathodal tDCS sessions, subjects will receive stimulation for 20 minutes with a current of 2.0 mA using a 5x5 cm electrode. During sham tDCS, a 2.0 mA current will be delivered for approximately 30 seconds before being extinguished over a course of seconds. The participant will complete pre/post language testing at each session in order to determine if the subject is a tDCS responder and if so, which site produces the best transient language improvement in that individual. Subjects who do not respond to tDCS will not be invited to move forward to the treatment phase.
  Interventions: Device: Transcranial Direct Current Stimulation (tDCS)
- Real tDCS (Active Comparator): Half of our tDCS responders will be randomized to a group receiving 10 sessions (divided in to two five-day periods) of real tDCS. During real tDCS sessions, subjects will receive stimulation for 20 minutes at a current of 2.0 mA with a 5x5 cm electrode at their optimal responder site previously determined.
  Interventions: Device: Transcranial Direct Current Stimulation (tDCS)
- Sham tDCS (Sham Comparator): Half of our tDCS responders will be randomized to a group receiving 10 sessions (divided in to two five-day periods) of sham tDCS. During sham tDCS, a 2.0 mA current will be delivered for approximately 30 seconds at the beginning of the sham condition before being extinguished over the course of seconds. Individuals randomized into the sham arm will be offered the option to crossover to real tDCS after their participation is complete.
  Interventions: Device: Transcranial Direct Current Stimulation (tDCS)

INTERVENTIONS:
Device: Transcranial Direct Current Stimulation (tDCS) — Transcranial direct current stimulation (tDCS) is a form of non-invasive neuromodulation that uses constant, low (1-2mA), direct current delivered via electrodes on the head.

SUMMARY:
This study proposes to use transcranial direct current stimulation (tDCS) in patients with chronic strokes and aphasia in order to characterize and enhance the mechanisms of language recovery following injury. Prior to enrollment subjects will undergo six "site-finding' sessions involving various placements of positively charged (anodal), negatively charged (cathodal), and sham stimulation over the damaged and intact hemispheres of the brain, along with standard tests of language. Subjects who are found to experience a transient improvement in language ability in this initial experiment will participate in an incomplete cross-over design study to determine if 10 sessions of tDCS stimulation lead to prolonged language benefit when delivered to the hemisphere and at the polarity shown previously to respond best to stimulation.

DETAILED DESCRIPTION:
Transcranial Direct Current Stimulation (tDCS) uses a small (typically 1-2 mA) electrical current which is passed through the scalp and is delivered for up to 20 minutes. Due to the safety and tolerability of tDCS, as well as its demonstrated capacity to temporarily enhance cognitive, motor and affective functions of the brain, there has been an explosion of interest in the technique since the first reports in 2000. tDCS has been used safely in a wide variety of domains including studies of the visual system, working memory, verbal fluency and motor function. tDCS has also been used safely to enhance brain function in subjects with a variety of brain pathologies including stroke, depression and Alzheimers Disease. In this study, the investigators hope to address whether tDCS can be used to enhance language function in individuals with post-stroke aphasia.

This two part experiment will address 1) Can tDCS lead to transient improvement in language ability in individuals with stroke and chronic aphasia? and 2) Does repeated tDCS lead to prolonged improved language ability in individuals with stroke and chronic aphasia?

In Experiment 1, which will be referred to as the 'site-finding' portion of this protocol, participants will undergo anodal, cathodal, and sham stimulation of the intact or injured hemisphere to determine what area of the brain responds best to tDCS. There will be six separate sessions which are spaced apart by at least 2 days. Tests of language will be used to characterize changes in performance that are induced in each condition.

In Experiment 2, subjects who had participated in Experiment 1 and were found to experience a transient improvement in language ability after receiving tDCS will participate. Subjects will be stimulated using the best montage from Experiment 1. This is an incomplete cross-over design study to determine if 10 sessions of tDCS stimulation delivered to the brain will lead to improvement in language. Improvement will be operationally defined as performance on one or more language measures that is significantly better than baseline and sham performance (i.e. non-stimulation conditions). Half of our subjects will be randomized to a group receiving 10 sessions (divided in to two five-day periods) of real tDCS. The other half of our subjects will be randomized to undergo sham stimulation before undergoing optional real tDCS stimulation. All subjects will engage in language rehearsal during stimulation. Tests of language will be used to characterize changes in performance that are induced by real and sham stimulation. Follow-up language testing will be performed at 2 weeks and 2 months after stimulation to determine whether tDCS can have prolonged effects on language.

ELIGIBILITY:
Inclusion Criteria:

* 1. Presence of aphasia attributable to one or more unilateral left hemispheric stroke(s)
* 2. The most recent stroke must have occurred 6 months prior to inclusion in the study
* 3. Must speak English as a native language
* 4. Must be able to understand the nature of the study, and give informed consent

Exclusion Criteria:

* 1. Subjects with bilateral strokes.
* 2. History of neurologic illness(es) other than stroke
* 3. Current unstable medical illness(es)
* 4. Epilepsy or Seizure(s) within the last six months
* 5. Subjects with metallic objects in the face or head other than dental apparatus such as braces, fillings, and implants.
* 6. Subjects with Pacemakers or ICDs
* 7. Diagnosed psychiatric disorders
* 8. Pregnancy
* 9. Current alcohol or drug abuse

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2010-07 (Actual); Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Change in naming ability after tDCS at different brain areas | 2 weeks
  We will contrast naming ability before and after daily tDCS at 5 different brain regions. A change in naming ability as a function of tDCS to a specific brain region will be taken as evidence that stimulation of that brain region is relevant to the performance of the behavioral task in question.
Change in overall aphasia severity after tDCS treatment | Through study completion, about 2 months
  We will contrast overall aphasia severity before and after tDCS comparing real vs. sham stimulation. A decrease in aphasia severity which is greater at real stimulation vs. sham stimulation suggests that tDCS may be a viable tool to improving language in post-stroke aphasia.